CLINICAL TRIAL: NCT06378112
Title: Extraction Socket Augmentation Using GTO vs. Apatos. A Randomized Controlled Clinical Study
Brief Title: Extraction Socket Augmentation. A Clinical Study
Acronym: GTO
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Universidad de Granada (Other)
Responsible Party: Principal Investigator, Manuel Toledano, Professor, Universidad de Granada
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2734/CEIH/2022
Record Dates: First submitted 2024-04-17; First posted 2024-04-22 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: Edentulous Alveolar Ridge With Labial Resorption
Keywords: Bone; Regeneration; Alveolar; Biomaterial

STUDY DESIGN:
Intervention Model Description: * Group 1 (test group): Guided bone regeneration procedure with GTO® as bone graft and soft collagenated cortical membrane (OsteoBiol® Lamina; Tecnoss srl) as graft stabilizer.
  * Group 2 (control): Guided bone regeneration procedure with Apatos Mix® cortico-cancellous heterologous bone mix (OsteoBiol®; Tecnoss srl) as bone graft and soft collagenated cortical membrane (OsteoBiol® Lamina; Tecnoss srl) as graft stabilizer.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1 (test group) (Experimental): Guided bone regeneration procedure with GTO® as bone graft and soft collagenated cortical membrane (OsteoBiol® Lamina; Tecnoss srl) as graft stabilizer.
  Interventions: Drug: GTO®
- Group 2 (control) (Active Comparator): Guided bone regeneration procedure with Apatos Mix® cortico-cancellous heterologous bone mix (OsteoBiol®; Tecnoss srl) as bone graft and soft collagenated cortical membrane (OsteoBiol® Lamina; Tecnoss srl) as graft stabilizer.
  Interventions: Drug: GTO®

INTERVENTIONS:
Drug: GTO® — After teeth extraction, a guided bone regeneration procedure will be performed using a bone graft and a soft collagenated cortical membrane as graft stabilizer. Implant placement surgery will also be performed.
  Other Names: Apatos®

SUMMARY:
Extraction socket preservation is defined as alveolar ridge preservation within the bone envelope remaining after tooth extraction, meanwhile ridge augmentation is defined as increasing the volume of alveolar ridge beyond the bony envelope at the time of tooth extraction. It is recommended to use in cases where extraction socket anatomy is intact. In contrast definition "extraction socket augmentation" defines alveolar ridge restoration when bony walls of the socket are partly or completely lost. In the case of severe loss (> 50%) of the buccal bone plate, preservation of hard tissue with a prolonged healing time before implant placement has been suggested.

The null hypothesis of this experimental work states that: (i) the two different bone graft materials gained the same amount of bone following horizontal ridge augmentation procedure; (i) the two different bone graft materials exhibit similar histological and histomorphometric results Therefore, the main purpose of the current study is to compare two different biomaterials using guided bone regeneration procedures in the ridge preservation/ augmentation (hard-tissue preservation).

DETAILED DESCRIPTION:
Patients needing teeth extraction and unitary implant placement will be recruited at the Dental School of the University of Granada (Máster de Cirugía Bucal).

Two study groups will be stated:

* Group 1 (test group): Guided bone regeneration procedure with GTO® as bone graft and soft collagenated cortical membrane (OsteoBiol® Lamina; Tecnoss srl) as graft stabilizer.
* Group 2 (control): Guided bone regeneration procedure with Apatos Mix® cortico-cancellous heterologous bone mix (OsteoBiol®; Tecnoss srl) as bone graft and soft collagenated cortical membrane (OsteoBiol® Lamina; Tecnoss srl) as graft stabilizer.

All employed Materials are commercially available and are completely approved to be used in humans. They are currently being used in dental practice in Europe, U.S.A. and many other countries. Eurofins Product Testing Italy S.r.l certifies that the manufacturer's full quality assurance system is compliant with Annex II of 93/42/EEC Medical Devices Directive and subsequent amenaments and upgrades (Certificate No. EPT0477.MDD.19/3209.1).

ELIGIBILITY:
Inclusion Criteria:

* Age: ≥ 18 years.

  * Good general health.
  * Single-tooth implant treatment. Presence of adjacent teeth and opposing occluding teeth (for measurement stent indexing).
  * Incisors, canines and premolars.
  * Presence of three intact socket walls after tooth extraction with a defect of more than 50% loss of the buccal ridge wall and no fragment of root should be left.
  * Reasons for tooth extraction: carious lesion, endodontic complication, root fracture and prosthetic reason.
  * Good oral and periodontal health.
  * Full-mouth plaque and bleeding < 20%.
  * Able and willing to follow study procedures and instructions.
  * Informed consent.

Exclusion Criteria:

* ≤ 18 years.

  * Comprised health. Existence of any systemic condition such as uncontrolled diabetes mellitus, cancer, HIV, disorders that compromise wound healing, chronic high dose steroid therapy, intravenous and oral bisphosphonate therapy, bone metabolic diseases, history of irradiation of the head and neck area, or any other immunosuppressive therapy that would contraindicate oral surgical treatment.
  * Absence of any adjacent teeth or the opposing occluding teeth.
  * Molars.
  * More than one bone wall defect.
  * Sinus pathology.
  * Allergy or hypersensitivity to medications or any of the products used throughout the study.
  * Heavy smokers (defined as >10 cigarettes per day or >1 cigar per day) or chew tobacco, including within 3 months prior to enrollment.
  * Untreated periodontitis.
  * Periapical or periodontal infection.
  * Full-mouth plaque and bleeding > 20%.
  * No informed consent

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-05-20 (Actual); Primary Completion 2025-01-15 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Dimensional bone changes | 3, 6 and 9 months
  Cone Beam Computed Tomography (CBCT) scans will be performed to each patient to evaluate the dimensional bone changes (height and width): one scan will be made immediately after regenerative surgery, and a second scan will be performed after a postoperative healing period of 6 months (prior to implant placement). Dimensional bone changes will be assessed superimposing and aligning the T0 (after regenerative surgery) and T1 (before implant placement).

CONTACTS AND LOCATIONS:
Overall Officials: Manuel Toledano, Professor, Principal Investigator — Universidad de Granada
Locations (1):
- Dental School, Granada, Spain

IPD SHARING:
Plan to Share IPD: Undecided